CLINICAL TRIAL: NCT02293174
Title: TRC-NW400 Retinal Fundus Camera Image Evaluation and Instrument Comparison Protocol
Brief Title: Retinal Fundus Camera Evaluation
Status: Completed | Type: Observational
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Other Study IDs: TOPCON-003-2014
Record Dates: First submitted 2014-11-11; First posted 2014-11-18 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Normal Healthy Subjects With no Known Ocular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal Healthy Eyes: Willing and able subjects with normal and healthy eyes
  Interventions: Device: Topcon TRC-NW400; Device: TRC-NW8; Device: TRC-NW400; Device: Canon-CR2; Device: Zeiss Visucam PRO

INTERVENTIONS:
Device: Topcon TRC-NW400 — Retinal Fundus Camera
Device: TRC-NW8 — Retinal Fundus Camera
Device: TRC-NW400 — Retinal Fundus Camera
Device: Canon-CR2 — Retinal Fundus Camera
Device: Zeiss Visucam PRO — Retinal Fundus Camera

SUMMARY:
Establish a normal baseline setting configuration for image capture using the Topcon TRC-NW400 non-mydriatic retinal camera.

DETAILED DESCRIPTION:
Establish a normal baseline setting configuration for image capture using the Topcon TRC-NW400 non-mydriatic retinal camera. While also comparing the images to other manufacturer's retinal cameras

ELIGIBILITY:
Inclusion Criteria:

* Subjects with no known ocular diseases

Exclusion Criteria:

* Subjects with known ocular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal subjects will be recruited from Topcon Medical Systems.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Fundus Image Grading | 1 Hour
  Determining the best display to reflect the real color of the retina

CONTACTS AND LOCATIONS:
Overall Officials: Danny Leung, Principal Investigator — Clinical Trial Manager
Locations (1):
- Topcon Medical Systems, Inc., Oakland, New Jersey, United States